CLINICAL TRIAL: NCT06883188
Title: A Pilot Randomised Study Comparing the Clinical Efficacy of Stopping Air Leak by Talc Pleurodesis or Autologous Blood Patch Therapy in Secondary Spontaneous Pneumothorax
Brief Title: Stop Air Leak by Talc or Autologous Blood Patch Therapy
Acronym: STOP
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Ka Pang Chan, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STOP
Record Dates: First submitted 2025-03-08; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Pneumothorax Spontaneous Secondary
Keywords: Persistent air leak; talc pleurodesis; autologous blood patch therapy
MeSH Terms: interventions — Dimethyl Sulfoxide

STUDY DESIGN:
Intervention Model Description: This is a single-centre, two-arm, open-label, randomized controlled trial including patients with spontaneous secondary pneumothorax and persistent air leak. Eligible patients will be randomised in a 1:1 ratio to receive either intrapleural administration of talc or autologous blood patch therapy. The digitalised air leak rate will be monitored continuously from randomisation till the removal of chest drain. Important endpoints include the rate of successful chest drain removal and reduction in air leak within 5 days after intrapleural intervention. This study will follow patients through their hospital stay and outpatient visits at 30 and 90 days after randomisation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- talc pleurodesis (Experimental): intrapleural instillation of talc slurry
  Interventions: Drug: talc powder
- Autolougs blood patch therapy (ABPT) (Active Comparator): intrapleural instillation of patient's venous blood
  Interventions: Biological: patient's own venous blood

INTERVENTIONS:
Drug: talc powder — intrapleural instillation of talc slurry
  Arms: talc pleurodesis
Biological: patient's own venous blood — intrapleural instillation of patient's own venous blood
  Arms: Autolougs blood patch therapy (ABPT)

SUMMARY:
Objectives: To compare the therapeutic efficacy and safety profiles of intrapleural talc pleurodesis versus autologous blood patch therapy(ABPT) in patients with secondary spontaneous pneumothorax(SSP) complicated by persistent air leak(PAL), and to assess the trial feasibility for a subsequent full-scale, multicentre randomised controlled trial(RCT).

Hypothesis: Talc pleurodesis and ABPT demonstrate comparable efficacy in stopping PAL and facilitating chest drain removal within 5 days.

Design and subjects: This single-centre, two-arm, open-label pilot RCT will recruit 30 patients with SSP and PAL persisting ≥5 days. Eligible patients will be randomised in a 1:1 ratio to receive intrapleural talc pleurodesis or ABPT. Digital chest drain systems will continuously record air leak rates from 24 hours before randomization until 120 hours post-intervention, ensuring objective, real-time data capture. Patients will be followed till 90 days post-discharge.

Interventions: Recruited subjects with PAL ≥5 days will be randomized in 1:1 ratio to receive talc pleurodesis or ABPT.

Main outcome measures: The primary outcome is complete cessation of air leak and successful chest drain removal within 5 days after the intervention. Secondary outcomes include absolute and percentage changes in digitally measured air leak rates, duration of chest drainage, recurrence of ipsilateral pneumothorax, need for additional pleural interventions, and safety outcomes such as drain blockage and pleural infection.

Data analysis and expected results: Data will be analysed on an intention-to-treat basis for all randomised subjects with regression models adjusting for confounders. The pilot outcomes will inform sample size calculations and refine design parameters for the proposed full-scale multicentre RCT.

DETAILED DESCRIPTION:
Pneumothorax, defined as the presence of air in the pleural space, is a common respiratory emergency that often necessitates prolonged hospitalisation. In cases where pneumothorax occurs in the setting of underlying chronic lung diseases (secondary spontaneous pneumothorax, SSP), the clinical course is considerably more severe. SSP patients are typically more hypoxic, more likely to develop persistent air leak (PAL) (exceeding 5-7 days), and experience longer hospital stays with higher in-patient mortality compared to those with primary spontaneous pneumothorax (PSP).

The management of SSP with PAL remains controversial despite its clinical significance. Numerous strategies, including chemical pleurodesis, autologous blood patch therapy (ABPT), implantation of endobronchial valves (EBV), and surgical pleurodesis, are employed in practice. However, many SSP patients are unsuitable for invasive procedures such as EBV placement or surgery, owing to their poor premorbid status. In this context, ABPT and chemical pleurodesis (often using talc) emerge as low-cost, bedside alternatives. Yet, current practices vary widely, and a lack of robust comparative evidence has left clinicians with no definitive guidance regarding the optimal management approach.

Talc pleurodesis, involving the intrapleural instillation of sterile talc powder, is a commonly adopted treatment for SSP with PAL. Retrospective studies indicate that 37.2% to 44.5% of SSP patients undergo chemical pleurodesis, with talc being the predominant agent. Reported treatment success is around 70%, with a median drainage duration of 12 days post-procedure. Adverse events, most notably chest pain affecting roughly one-third of patients, are not uncommon, although more serious complications such as respiratory distress occur in only 1.6% of cases. Nonetheless, these findings are derived from studies with retrospective designs and variable methodologies, limiting firm conclusions on efficacy and safety.

In contrast, ABPT has been proposed as a promising alternative for managing PAL. This technique involves the intrapleural instillation of autologous blood with the aim of sealing the air leak, initially developed for PAL in post-operative pneumothorax. Several small-scale retrospective and prospective studies have suggested that ABPT can achieve cessation in 26% to 91% of cases, with some reports showing 71.7% to 84.0% of patients experiencing complete resolution within five days. Moreover, ABPT appears safe for repeated administration, with adverse events reported at incidences ranging from 0% to 16%. However, the heterogeneous outcomes likely reflect differences in blood dosage, timing of intervention, number of administrations, and varying definitions of PAL among studies.

Given the controversy and the limitations of existing evidence, a multicentre randomised controlled trial (RCT) comparing talc pleurodesis with ABPT is imperative. To achieve this, a pilot study is designed to rigorously address methodological weaknesses by standardising the timing of pleural interventions, employing a digital chest drain system for precise, quantitative measurement of air leak, and adopting unified criteria for treatment success.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Radiographically proven pneumothorax and underlying lung disease (either pre-existing or shown in diagnostic imaging at presentation)
* Spontaneous onset of pneumothorax, not related to trauma or iatrogenic procedure
* SSP with air leak persists for ≥3 days after the first radiographic evidence of pneumothorax
* Intend to administer talc or autologous blood patch therapy (ABPT) to stop the air leak as the next step of treatment

Exclusion Criteria:

* A chest drain size smaller than Fr 12
* Bilateral pneumothorax
* Impaired blood clotting, including baseline INR > 1.5, platelet < 150 x 10^9/L, use of therapeutic dose anticoagulant or dual-antiplatelet agents
* Active or recent (within 6 weeks) pleural infection
* Septicaemia or active extrapleural infection (e.g. pneumonia)
* Use of long-term systemic corticosteroids or immunosuppressant
* Previously received talc or ABPT to the ipsilateral pleural space for the current episode of pneumothorax
* Known sensitivity to talc
* Has had a previous pneumonectomy (either on the same or contralateral side)
* Patients who are pregnant or lactating (females of childbearing potential must have a negative pregnancy test before randomisation)
* Expected survival of less than three months from a different pathology to this pneumothorax (e.g. metastatic malignancy)
* Cognitively impaired and physically unable to follow the turning procedure during intrapleural procedure, or at risk of self-removing chest drain
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Complete cessation of air leak within 5 days of study intervention | 5 days
  Complete cessation of air leak for more than 24 hours and successful chest drain removal within 5 days after talc pleurodesis or ABPT

SECONDARY OUTCOMES:
Change in the average rate of air leak | 5 days
  Absolute reduction and percentage change in the average rate of air leak (in mL/min) from randomisation to 5 days after the study interventions
Time to air leak cessation | 30 days
  Time from study intervention to complete cessation of air leak and successful removal of all chest drain(s) (in hours)
Length of hospital stay | 3 months
  Length of hospital stay after study intervention (in days)
Recurrence of pneumothorax | 3 months
  Recurrence of ipsilateral pneumothorax after study intervention
Number of patients requiring additional intervention | 3 months
  The need for additional (unplanned or elective) interventions for persistent air leak, which includes needle aspiration, chest drain insertion, implantation of endobronchial valve, surgery
Pain score | 5 days
  Pain score in visual analogue scale, score ranges from 0 to 10, with 0 means no pain, and 10 means the worst pain ever
Breathlessness score | 5 days
  Breathlessness by visual analogue scale, score ranges from 0 to 100, with 0 means no breathlessness, and 100 means the worst breathlessness ever
Adverse events | 3 months
  Occurrence of adverse events directly related to study interventions (e.g. drain blockage, pleural infection / empyema, fever, acute respiratory distress syndrome)
Spirometry parameter | 3 months
  Pre-bronchodilater spirometry parameters (forced expiratory volume in 1 second and forced vital capacity, both in liter) at 1 and 3 month follow up
6-minute walking distance | 3 months
  6-minute walking distance (in meter) at 1 and 3 month follow up

CONTACTS AND LOCATIONS:
Overall Officials: David SC Hui, MD, Study Director — Chinese University of Hong Kong

IPD SHARING:
Plan to Share IPD: No